CLINICAL TRIAL: NCT00528463
Title: a Prospective Case Series of Pre-emptive Pre-amputation Sciatic Nerve Block to Prevent Lower Limb Phantom Pain
Brief Title: Pre-emptive Sciatic Bloc to Prevent Lower Limb Phantom Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Étienne de Médicis, CHUS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: edm1
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2007-09

CONDITIONS: Phantom Limb Pain
Keywords: Pre-emptive analgesia; Peripheral nerve block (sciatic); phantom lomb pain
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sciatic block (Experimental): One arm, all patient studied received a block
  Interventions: Procedure: sciatic nerve block

INTERVENTIONS:
Procedure: sciatic nerve block — Sciatic nerve block, Labatt approach, with a stimuplex needle and catheter. Once localized, a bolus of 20 mL ropivacaine 1,0% is given through the catheter and is followed by a perfusion of ropivacaine 0,2% 6-10 mL/hre for at least 24 hours pre-op and 48 hours post-op

SUMMARY:
Phantom limb pain is a complication of amputation. Although pre-empitve epidural analgesia was once thought to prevent such a com plication, recent studies did not demonstrate this. Peripheral blocks are more powerful then epidurals, and can even influence somatotropic representation in the brain. This a prospective case series in which the investigators hope to show a decrease, against historical control, of the incidence of post-operative amputation lower limb phantom pain. The investigators established the block at least 24 hours pre-operative and continue it for at least 2 days. Patient are followed daily for the 1st 3 days and then up to 3 month for the incidence of phantom limb pain. The investigators hope to recruit 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for lower limb amputation

Exclusion Criteria:

* Inability to consent
* Contraindication to peripheral nerve block
* Inability to perform the block
* Inadequate time frame (less than 24 hours prior to surgery)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
incidence of lower limb phantom pain | 3 month post amputation

CONTACTS AND LOCATIONS:
Overall Officials: ETIENNE DE MEDICIS, MD, MSC, Principal Investigator — Université de Sherbrooke
Locations (1):
- CHU, Sherbrooke, Quebec, Canada